CLINICAL TRIAL: NCT07131488
Title: Research on the Mechanisms and Intervention Strategies for Physical Activity Promotion in Frail Patients With Cardiovascular-Kidney-Metabolic Syndrome From a Temporal Self-Regulation Perspective
Brief Title: Mechanisms and Interventions for Physical Activity in Frail Cardiovascular-kidney-metabolic Syndrome Patients: A Temporal Self-Regulation Approach
Acronym: CKM
Status: Not yet recruiting | Type: Observational
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Zhongmin Fu, Principal Investigator, Nanjing Medical University
Other Study IDs: 20250731
Record Dates: First submitted 2025-07-31; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Cardiovascular-kidney-metabolic Syndrome
Keywords: Time-limited Self-regulation Theory; physical activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Middle-aged frail population with CKM syndrome: This was a non-interventional longitudinal study，primarily focuses on the mechanisms and factors influencing physical activity in middle-aged CKM syndrome patients.

SUMMARY:
Longitudinal physical activity data and associated factors were collected at baseline (diagnosis), 3-month, 6-month, and 9-month follow-ups in cardiovascular-kidney-metabolic syndrome patients.

DETAILED DESCRIPTION:
This study targets the frail population with early-middle-age CKM syndrome. Grounded in the Time-limited Self-regulation Theory (TST), it employs behavioral data analysis, theoretical variable modeling, and intervention strategy development to systematically identify risk trajectories and influencing pathways of physical activity (PA) insufficiency, thereby formulating stratified and classified intervention strategies to enhance PA levels. The research comprises three key components:

Research Component 1: Risk Prediction Model for PA Insufficiency in Frail CKM Syndrome Patients Early-middle-age frail CKM syndrome patients exhibit significant PA insufficiency and behavioral variability at the disease onset. Early identification of PA evolution trends and high-risk groups is crucial for timely intervention and precise resource allocation.

Objective:

To determine "who is more likely to sustain PA insufficiency" by constructing a trajectory identification model and risk prediction tool using longitudinal data, analyzing dynamic PA behavior patterns, and quantifying multifactorial risk probabilities to support subsequent intervention mechanisms and strategy classification.

Study Design:

Exploring PA Trajectories in Frail CKM Syndrome Patients

Target Population: Early-middle-age frail CKM patients (aligned with AHA lifestyle management guidelines).

Method: Prospective longitudinal study with multi-timepoint data collection.

Analysis: Group-based trajectory modeling (GBTM) to delineate PA dynamics, identifying high-risk trends (e.g., persistent insufficiency, steep decline).

Developing a Risk Prediction Model for PA Insufficiency

Dependent Variable: PA trajectory classification (e.g., stable-high, persistent-low, fluctuating).

Predictors: Sociodemographics, health behaviors, and environmental factors.

Method: Multi-class machine learning (XGBoost) to identify key predictors and quantify risk probabilities.

Output: Interactive visualization tool for community-level screening of high-risk individuals.

Research Component 2: TST-Based Mechanisms of PA Promotion in Frail CKM Syndrome Patients

To elucidate the key determinants and moderators of PA insufficiency, this study leverages TST's six core variables:

Behavioral intention

Consistency beliefs

Self-control capacity

Delay discounting tendency

Environmental cue perception

Habit formation strength

Methodological Approach:

Dynamic Feature Engineering:

Multi-timepoint measurement of TST variables → Derived metrics (baseline level, trend, mean, variability).

Dimensionality Reduction:

LASSO regression + PCA to mitigate multicollinearity.

Predictive Modeling:

XGBoost classification (trajectory groups as outcomes) + SHAP analysis to rank variable contributions.

Causal Pathway Analysis:

Generalized structural equation modeling (GSEM) to identify mechanistic pathways.

Outcome:

Prioritized modifiable factors (e.g., self-control > environmental cues) for tailored interventions.

Research Component 3: TST-Driven PA Promotion Strategies for Frail CKM Syndrome Patients Goal: Translate mechanistic insights into actionable, precision strategies for behavior change.

Strategy Development Framework:

Intervention Targets:

Mechanistic variables (e.g., enhancing self-control in "persistent-low" trajectory patients).

Three Strategy Archetypes:

Intrinsic Motivation Modulation (e.g., goal-setting interventions)

Social Support Activation (e.g., peer coaching)

Environmental Cue Optimization (e.g., neighborhood walkability enhancements)

Strategy Prioritization:

Analytic Hierarchy Process (AHP) to weight strategies by feasibility, acceptability, and efficacy.

Deliverable:

A modular "PA Promotion Toolkit" for phased, adaptive community interventions.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥45 years and <60 years;

Frailty status assessed by Fried phenotype criteria, including those diagnosed with frailty or pre-frailty;

Meeting AHA guideline criteria for Stage 1-2 CKM syndrome (diagnostic details in Table 1);

Ability to communicate normally and use smartphones or wearable devices;

Willingness to participate in surveys and follow-up;

Additional Note on PREVENT Equation:

The PREVENT equation, developed by the American Heart Association (AHA), is a cardiovascular disease (CVD) risk prediction tool. It calculates 10-year CVD risk based on:

Age, sex

Total cholesterol, HDL-C

Systolic blood pressure, BMI

eGFR

History of diabetes, smoking

Use of antihypertensive or lipid-lowering medications

Exclusion Criteria:

* Severe cognitive impairment (e.g., MMSE score <10 or clinical dementia diagnosis);

Severe psychiatric/psychological disorders (e.g., schizophrenia, major depressive disorder with suicidal ideation);

Advanced chronic diseases including:

End-stage renal disease (eGFR <15 mL/min/1.73m² or on dialysis)

Metastatic cancer (stage IV per AJCC criteria)

Cardiorespiratory insufficiency (NYHA Class III-IV heart failure or COPD GOLD Stage D)

Severe osteoarthritis (Kellgren-Lawrence Grade 4 with functional limitation)

Major surgery or acute illness within 3 months (e.g., myocardial infarction, stroke, or major trauma requiring hospitalization);

Physical disabilities impairing mobility (e.g., amputation, paralysis, or severe Parkinsonism with Hoehn & Yahr Stage ≥3).

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study was conducted at the First Affiliated Hospital of Nanjing Medical University (Jiangsu Province Hospital), enrolling 614 middle-aged adults with frailty and cardiovascular-kidney-metabolic (CKM) syndrome. Participants who met the inclusion/exclusion criteria and provided written informed consent were prospectively followed for 12 months.
Sampling Method: Non-Probability Sample
Enrollment: 614 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2026-10-12 (Estimated); Study Completion 2026-10-12 (Estimated)

PRIMARY OUTCOMES:
Consideration of Future Consequences Scale (CFC-S) | Baseline , 3 months, 6 months, 9 months
  The Consideration of Future Consequences Scale (CFC-S), developed by Strathman et al., includes two dimensions: consideration of the present (items 3, 4, 5, 9, 10, 11, 12) and consideration of the future (items 1, 2, 6, 7, 8). The Chinese version was cross-culturally adapted by Feng Jiaxi et al. The scale includes 12 items, rated on a 7-point Likert scale, where 1 means "not at all like me" and 7 means "exactly like me." Internal consistency coefficients in elderly populations are 0.71 and 0.80 for the two dimensions, and split-half reliability is 0.69 and 0.78, indicating good psychometric properties.
Global Physical Activity Questionnaire (GPAQ) | Baseline , 3 months, 6 months, 9 months
  It includes four domains: work, transportation, recreation, and sedentary behavior. The questionnaire assesses the participant's PA in these four areas over the course of a week. PA in the work and recreation domains is further classified into vigorous and moderate levels. The questionnaire contains 16 items, and only activities lasting more than 10 minutes are considered relevant PA.The higher the activity intensity, the greater the MET value, meaning the body consumes more energy. High PA Level: At least three days of vigorous-intensity activity per week, with a total MET value of at least 1500 METs, or daily moderate-to-vigorous activity with a total MET value of at least 3000 METs per week.
  Moderate PA Level: At least three days of vigorous-intensity activity per week.Low PA Level: Insufficient activity, where the individual does not meet the moderate-to-vigorous intensity activity standard.

SECONDARY OUTCOMES:
Monetary Choice Questionnaire (MCQ) | Baseline , 3 months, 6 months, 9 months
  he Monetary Choice Questionnaire (MCQ), developed by Kirby et al., is a widely validated tool to assess delay discounting. An Excel-based tool for automatic calculation of discount rates is available for free.
Exercise Benefits/Barriers Scale (EBBS) | Baseline , 3 months, 6 months, 9 months
  The Exercise Benefits/Barriers Scale (EBBS) measures perceived exercise benefits and barriers in CKM syndrome patients. Higher scores indicate greater perception of exercise benefits and fewer barriers.
Intentions | Baseline , 3 months, 6 months, 9 months
  Participants are informed of the recommended weekly PA levels: 150 minutes of moderate-intensity aerobic exercise or 75 minutes of vigorous-intensity aerobic exercise, plus at least two days of muscle-strengthening exercises. Physical activity intentions will be measured using a subscale from the TPB questionnaire, developed and validated by Ajzen (1991) and adapted for China by Hu et al. (2008). Intention is assessed using three items on a scale from 1 (strongly disagree) to 6 (strongly agree). Higher average scores indicate stronger intentions. This subscale has excellent reliability, with a Cronbach's α of 0.944.
Self-Report Habit Index (SRHI) | Baseline , 3 months, 6 months, 9 months
  The Self-Report Habit Index (SRHI), a commonly used measure of habits, consists of 12 items covering three dimensions: behavioral repetition history, lack of awareness, and lack of control. The behavior X (defined as moderate-to-vigorous physical activity in this study) is assessed by participants through these 12 items. A 5-point Likert scale is used in the Chinese version, which has a Cronbach's α of 0.961.
Healthy Neighborhood Survey for Community-Dwelling Older Adults | Baseline , 3 months, 6 months, 9 months
  The community leisure environment is assessed in terms of 10 aspects: interesting architecture, clean and tidy surroundings, attractive environment, easy walkability, suitability for walking, abundant trees, availability of exercise opportunities, sufficient exercise facilities, ability to attract residents to walk, and ability to encourage residents to exercise. The scale ranges from 1 to 5, with options for "Strongly Disagree," "Disagree," "Neutral," "Agree," and "Strongly Agree," reflecting the respondent's recognition of various aspects of the community leisure environment.
Brief Self-Control Scale (BSCS) | Baseline , 3 months, 6 months, 9 months
  Self-control, an important aspect of self-regulation, will be measured using the Brief Self-Control Scale (BSCS), originally developed by Morean et al. The scale consists of 7 items measuring two dimensions: self-discipline (items 1, 3, 5) and impulse control (items 2, 4, 6, 7). Higher scores indicate better self-regulation. The Chinese version of the BSCS has a Cronbach's α of 0.83.
Multidimensional Frailty | baseline
  Multidimensional frailty is assessed based on the Frailty Integration Model and the Tilburg Frailty Indicator. The indicators include physical frailty, psychological frailty, and social frailty. Frailty is measured by calculating a total frailty score, with a maximum score of 15 points. A score of ≥5 indicates multidimensional frailty, with higher scores indicating greater severity of frailty.
  Physical Frailty: The maximum score is 8 points, with ≥3 points indicating physical frailty.
  Psychological Frailty: The maximum score is 4 points, with ≥1.5 points indicating psychological frailty.
  Social Frailty: The maximum score is 3 points, with ≥1.5 points indicating social frailty
Charlson Comorbidity Index (CCI) | baseline
  The CCI evaluates comorbidities and disease severity, with a higher score indicating greater comorbidity. Different diseases have different weightings, and the index has been updated to include 23 diseases, including hypertension, depression, and the use of anticoagulants. The higher the score, the more severe the comorbidities.

IPD SHARING:
Plan to Share IPD: No